CLINICAL TRIAL: NCT00693927
Title: Nonmyeloablative Stem Cell Transplantation With CD8-depleted or Unmanipulated Peripheral Blood Stem Cells: A Prospective Randomized Phase II Trial
Brief Title: Nonmyeloablative Stem Cell Transplantation With CD8-depleted or Unmanipulated Peripheral Blood Stem Cells (PBSC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Yves Beguin, Prof, University of Liege
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Minitransplant - random
Record Dates: First submitted 2008-05-29; First posted 2008-06-09 (Estimated); Last update posted 2011-09-02 (Estimated); Status verified 2011-09

CONDITIONS: Hematologic Malignancies
Keywords: Hematopoietic cell transplantation; Allogeneic; Nonmyeloablative; CD8-depletion; PBSC; GVHD; Hematological malignancies and renal cell carcinoma
MeSH Terms: conditions — Hematologic Neoplasms; Carcinoma, Renal Cell | interventions — Transplantation Conditioning

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Unmanipulated PBSC
  Interventions: Procedure: Unmanipulated PBSC after nonmyeloablative conditioning
- 2 (Experimental): CD8-Depleted PBSC
  Interventions: Procedure: CD8-depleted PBSC after nonmyeloablative conditioning

INTERVENTIONS:
Procedure: Unmanipulated PBSC after nonmyeloablative conditioning — Conditioning regimen with 2 Gy TBI with or without added fludarabine (90 mg/m2).
  Unmanipulated PBSC from HLA-identical sibling or HLA-matched related or unrelated donor
  Arms: 1
Procedure: CD8-depleted PBSC after nonmyeloablative conditioning
  Other Names: Conditioning regimen with 2 Gy TBI with or without added fludarabine (90 mg/m2).; CD8-depleted PBSC from HLA-identical sibling or HLA-matched related or unrelated donor
  Arms: 2

SUMMARY:
Prospective randomized study of allogeneic minitransplantation from HLA-identical family or unrelated donors comparing unmanipulated or CD8-depleted PBSC. The conditioning regimen will be 2 Gy TBI alone (related donor with low-risk of transplant rejection) or 2 Gy TBI and 3 x 30 mg/m2 fludarabine (unrelated donor or high risk of transplant rejection). Patients will receive a short but intensive immunosuppressive treatment (cyclosporine and mycophenolate mofetil) to ensure both graft-versus-host and host-versus-graft tolerance. The rationale for using PBSC instead of marrow transplant is to avoid general anesthesia of the donor and to minimize the risk of rejection. The rationale for CD8+ depletion is to diminish the risk of GVHD after PBSC transplantation or DLI.

ELIGIBILITY:
1. Patients

   1.1. Diseases

   Malignant diseases confirmed histologically and not rapidly progressing:
   * Hematologic malignancies
   * AML;
   * ALL;
   * CML and other myeloproliferative disorders;
   * MDS;
   * Multiple myeloma;
   * CLL;
   * Non-Hodgkin's lymphoma;
   * Hodgkin's disease.
   * Non-hematologic malignancies
   * Renal cell carcinoma (metastatic).

   1.2. Inclusion criteria
   * Male or female; female patients must use a reliable contraception method;
   * Age lower than 70 yrs (family donor) or lower than 65 yrs (unrelated donor);
   * HIV negative;
   * No terminal organ failure;
   * No uncontrolled infection, arrhythmia or hypertension;
   * Family donor (HLA-identical) or unrelated donor (matched for A-B by low resolution typing and for DRB1-DQB1 by high resolution typing);
   * No previous radiation therapy precluding the use of 2 Gy TBI
   * Informed consent given by patient or his/her guardian if of minor age.

   1.3. Clinical situations
   * Theoretical disease indication for a standard allo-transplant, but not feasible because:
   * Age > 55 yrs;
   * Unacceptable end organ performance;
   * Patient's refusal.
   * Indication for a standard auto-transplant:

     * perform mini-allotransplantation 2-6 months after standard autotransplant.
   * Not an indication for intensification but a potential candidate for cellular immunotherapy.
2. Donors

2.1. Inclusion criteria

* Related to the recipient (sibling, parent or child) or unrelated;
* Male or female;
* Weight > 15 Kg (because of leukapheresis);
* HIV negative;
* No major contraindication for allogeneic PBSC donation by generally accepted criteria;
* Informed consent given by donor or his/her guardian if of minor age.

2.2. Exclusion criteria

* Any condition not fulfilling inclusion criteria;
* Unable to undergo leukapheresis because of poor vein access or other reasons.

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2002-03; Primary Completion 2005-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Incidence of acute GVHD in CD8-depleted versus unmanipulated groups | 180 days
Incidence of chronic GVHD (overall and extensive) in CD8-depleted versus unmanipulated groups. | 1-year

SECONDARY OUTCOMES:
Incidence of graft rejection [according to the risk of transplant rejection (see table 1 above)] in CD8-depleted versus unmanipulated groups. | 1-year
T cell (CD3) and myeloid (CD13) chimerism in CD8-depleted versus unmanipulated groups. | 1-year and then long term
Quality and timing of immune reconstitution in CD8-depleted versus unmanipulated groups. | 1-year

CONTACTS AND LOCATIONS:
Overall Officials: Yves Beguin, MD, PhD, Study Chair — University of Liege
Locations (1):
- CHU Sart Tilman, Liège, Liege, Belgium